CLINICAL TRIAL: NCT04832321
Title: Measuring Beliefs and Norms About Persons With Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Alexander Tsai, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2013P000395_1
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Stigma
MeSH Terms: conditions — Alcoholism; Social Stigma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Study participants are randomly assigned to be read vignettes with slight changes in wording. Neither study participants nor outcomes assessors are provided with information about "treatment" assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- No intervention: V1: Control (No Intervention): This version of the survey questionnaire depicts a young man with no symptoms of alcohol use disorder
- Experimental: V2: Alcohol Use Disorder (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young man with symptomatic, untreated alcohol use disorder.
  Interventions: Other: Survey questionnaire
- Experimental: V3: Alcohol Use Disorder + Treatment with Response (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young man with symptomatic, untreated alcohol use disorder who is successfully treated with complete response.
  Interventions: Other: Survey questionnaire
- Experimental: V4: Alcohol Use Disorder + Treatment with Relapse (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young man with symptomatic, untreated alcohol use disorder who is successfully treated with partial relapse.
  Interventions: Other: Survey questionnaire
- Experimental: V5: Alcohol Use Disorder + Economic Impact (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young man with symptomatic, untreated alcohol use disorder whose untreated alcohol use disorder negatively affects his family's finances.
  Interventions: Other: Survey questionnaire
- Experimental: V6: Alcohol Use Disorder + Economic Impact + Treatment with Response (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young man with symptomatic, untreated alcohol use disorder whose untreated alcohol use disorder negatively affects his family's finances, who is then successfully treated with complete response.
  Interventions: Other: Survey questionnaire
- Experimental: V7: Alcohol Use Disorder + Economic Impact + Treatment with Relapse (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young man with symptomatic, untreated alcohol use disorder whose untreated alcohol use disorder negatively affects his family's finances, who is then successfully treated with partial relapse and continued negative economic impact.
  Interventions: Other: Survey questionnaire

INTERVENTIONS:
Other: Survey questionnaire — Each version of the questionnaire portrays a young Ugandan man with different profiles of illness severity, treatment, and treatment response.
  Arms: Experimental: V2: Alcohol Use Disorder; Experimental: V3: Alcohol Use Disorder + Treatment with Response; Experimental: V4: Alcohol Use Disorder + Treatment with Relapse; Experimental: V5: Alcohol Use Disorder + Economic Impact; Experimental: V6: Alcohol Use Disorder + Economic Impact + Treatment with Response; Experimental: V7: Alcohol Use Disorder + Economic Impact + Treatment with Relapse

SUMMARY:
Survey experiment to estimate drivers of stigma toward people with alcohol use disorder

DETAILED DESCRIPTION:
Despite significant advances in scientific understanding of substance use disorders accompanied by significant advances in treatment and improvements in prognosis, substance use disorder remains highly stigmatized throughout the world. Previous studies suggest that portraying alcohol use disorder as treatable can reduce negative attitudes toward persons with alcohol use disorder. This randomized controlled trial compares the effects of exposing study participants to vignettes portraying persons with untreated and symptomatic alcohol use disorder vs. treated alcohol use disorder with complete response vs. treated alcohol use disorder with relapse, with and without adverse economic impacts. It is hypothesized, based on prior work, that study participants exposed to vignettes depicting treated alcohol use disorder with completed response would have the greatest effect on reducing negative attitudes toward persons with alcohol use disorder, followed by treated alcohol use disorder with relapse and untreated and symptomatic alcohol use disorder, and that adverse economic impacts will exacerbate negative attitudes toward persons with alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

* All adults who consider Nyakabare their primary place of residence and who are capable of providing consent

Exclusion Criteria:

* Minors younger than 18 years of age, with the exception of emancipated minors
* Persons who do not consider Nyakabare Parish their primary place of residence, e.g., persons who happen to be visiting Nyakabare at the time of the survey or who own a home in Nyakabare but spend most of their time outside the parish
* Persons with psychosis, neurological damage, acute intoxication, or other cognitive impairment (all of which are determined informally in the field by non-clinical research staff in consultation with a supervisor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1363 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Social Distance | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate)
  Willingness to have the man portrayed in the vignette to marry into the study participant's family (single item, culturally adapted instrument developed specifically for this study; response options yes/no)
Perceived Norms about Social Distance | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate)
  Study participant's perception of the extent to which other people would be willing to have the man portrayed in the vignette to marry into their families (single item, culturally adapted instrument developed specifically for this study; response options on a Likert-type scale: 1=all or almost all; 2=more than half but less than all; 3=fewer than half but more than no one; 4=very few or no one)
Negative Attitudes (Attribution) | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate)
  Personal belief that the symptoms of the man portrayed in the vignette represent divine punishment (single item, culturally adapted instrument developed specifically for this study; response options yes/no)
Perceived Norms about Negative Attitudes (Attribution) | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate)
  Study participant's perception of the extent to which other people believe that the symptoms of the man portrayed in the vignette represent divine punishment (single item, culturally adapted instrument developed specifically for this study; response options on a Likert-type scale: 1=all or almost all; 2=more than half but less than all; 3=fewer than half but more than no one; 4=very few or no one)
Negative Attitudes (Shame) | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate)
  Personal belief that the symptoms of the man portrayed in the vignette bring shame upon his family (single item, culturally adapted instrument developed specifically for this study; response options yes/no)
Perceived Norms about Negative Attitudes (Shame) | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate)
  Study participant's perception of the extent to which other people believe that the symptoms of the man portrayed in the vignette bring shame upon his family (single item, culturally adapted instrument developed specifically for this study; response options on a Likert-type scale: 1=all or almost all; 2=more than half but less than all; 3=fewer than half but more than no one; 4=very few or no one)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Tsai, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No